CLINICAL TRIAL: NCT06976970
Title: Diet Quality And Metabolic Syndrome In Adult Individuals: Evaluation Of Turkey Nutrition And Health Survey 2017
Status: Active, not recruiting | Type: Observational
Sponsor: Elif Akbas (Other)
Responsible Party: Sponsor-Investigator, Elif Akbas, Research Assistant, Marmara University
Organization: Marmara University (Other)
Other Study IDs: OMÜ KAEK 2024/120
Record Dates: First submitted 2025-04-22; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Diet Quality; Healthy Eating Index (HEI-2015); Dietary Inflammatory Index (DII); Mediterranean Diet Score (mMDS); DASH Diet
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metabolic Syndrome group
- Non-Metabolic Syndrome group

SUMMARY:
This study investigates how the quality of a person's diet may be related to metabolic syndrome, which includes health issues such as high blood pressure, high blood sugar, and abdominal obesity. The research uses existing data from the 2017 Turkey Nutrition and Health Survey, focusing on adults aged 19 and over. The study does not involve any medical treatments or new data collection. It aims to support public health efforts by identifying links between eating patterns and metabolic health in the Turkish population.

DETAILED DESCRIPTION:
This study is a secondary analysis of the 2017 Turkey Nutrition and Health Survey (TNHS), which was conducted by the Ministry of Health to assess the health and nutritional status of the Turkish population. The objective of this cross-sectional observational study is to evaluate the relationship between diet quality and the presence of metabolic syndrome (MetS) among Turkish adults aged 19 years and older.

Diet quality will be assessed using several validated dietary indices, including the Healthy Eating Index-2015 (HEI-2015), the Dietary Inflammatory Index (DII), the modified Mediterranean Diet Score (MDS), and the DASH (Dietary Approaches to Stop Hypertension) score. These indices provide a comprehensive evaluation of overall dietary patterns and their potential impact on metabolic health.

Metabolic syndrome will be defined based on the Joint Interim Statement (2009) criteria. Participants will be classified as having metabolic syndrome if at least three of the following five components are present: abdominal obesity, elevated blood pressure or receiving antihypertensive treatment, reduced HDL cholesterol levels or receiving treatment for dyslipidemia, elevated triglyceride levels or receiving lipid-lowering therapy, and elevated fasting blood glucose or receiving treatment for hyperglycemia.

Statistical analysis will include descriptive statistics, t-tests or Mann-Whitney U tests for comparisons between MetS and non-MetS groups, and multivariate logistic regression analyses to determine the associations between dietary indices and the likelihood of having MetS, adjusting for relevant sociodemographic and lifestyle covariates.

Statistical analyses were conducted using SPSS version 22.0. Descriptive statistics included frequencies and percentages for categorical variables and means with standard deviations or medians with ranges for continuous variables, depending on the distribution. Normality was assessed using the Shapiro-Wilk test. Group comparisons were performed using the Mann-Whitney U test or Kruskal-Wallis test for non-normally distributed variables and the Chi-square test for categorical variables. Correlations between continuous variables were evaluated using Spearman's rank correlation coefficient. Binary logistic regression analysis was used to identify factors associated with the presence of metabolic syndrome. A p-value of <0.05 was considered statistically significant.

This study is expected to contribute to the national evidence base on dietary patterns and metabolic health and to inform public health strategies aiming to reduce the burden of non-communicable diseases in Turkiye.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older
* Participated in the 2017 Turkey Nutrition and Health Survey (TNHS)

Exclusion Criteria:

* Pregnant or lactating women, individuals with cancer, psychiatric or neurological disorders, those on specific therapeutic diets, individuals with missing key variables, and those with implausible energy intake levels (<800 or >4000 kcal/day for men, <500 or >3500 kcal/day for women).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 19 years and older who participated in the 2017 Turkey Nutrition and Health Survey (TNHS), conducted by the Turkish Ministry of Health. This secondary data analysis includes participants with complete dietary, demographic, anthropometric, and biochemical data. Exclusion criteria were: pregnant or lactating women, individuals with cancer, psychiatric or neurological disorders, those on specific therapeutic diets, individuals with missing key variables, and those with implausible energy intake levels (<800 or >4000 kcal/day for men, <500 or >3500 kcal/day for women).
Sampling Method: Probability Sample
Enrollment: 4915 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Metabolic Syndrome (MetS) | Day 1
  The primary outcome is the presence or absence of metabolic syndrome, defined according to the Joint Interim Statement criteria (2009). Participants are classified as having MetS if they meet at least three of the following five components: abdominal obesity, elevated blood pressure, elevated fasting glucose, elevated triglycerides, and reduced HDL cholesterol.
HEI-2015 Score | Day 1
  Diet quality will be assessed using the Healthy Eating Index-2015 (HEI-2015).
Dietary Inflammatory Index (DII) | Day 1
  Diet quality will be assessed using the Dietary Inflammatory Index (DII).
Mediterranean Diet Score (MDS) | Day 1
  Diet quality will be assessed using the Mediterranean Diet Score (MDS).
DASH Score (Dietary Approaches to Stop Hypertension) | Day 1
  Diet quality will be assessed using the DASH (Dietary Approaches to Stop Hypertension) score.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Akbas, Research Assistant, Principal Investigator — Marmara University; Yasemin Ertas Ozturk, Assistant Professor, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No